CLINICAL TRIAL: NCT02215967
Title: A Phase I Clinical Trial of T-Cells Targeting B-Cell Maturation Antigen for Previously Treated Multiple Myeloma
Brief Title: Study of T Cells Targeting B-Cell Maturation Antigen for Previously Treated Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Kochenderfer, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 140168; 14-C-0168
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Myeloma, Plasma-Cell; Myeloma-Multiple
Keywords: Immunotherapy; Anti-BCMA-CAR; Gene Therapy; Adoptive T Cell Therapy; Plasma Cell Malignancy
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; bis(3-bis(4-chlorophenyl)methyl-4-dimethylaminophenyl)amine; Receptors, Chimeric Antigen; Automobiles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Multiple Myeloma (Experimental): Dose Escalation with 5 dose levels based on the patients actual bodyweight
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Anti-B-cell maturation antigen (BCMA) chimeric antigen receptor (CAR) T cells

INTERVENTIONS:
Drug: Cyclophosphamide — 300 mg/m^2 intravenous (IV) over 30 minutes on days -5, -4, and -3
  Other Names: Cytoxan
Drug: Fludarabine — 30 mg/m^2 intravenous (IV) over 30 minutes immediately following the cyclophosphamide on day -5, -4, and -3
  Other Names: Fludara
Biological: Anti-B-cell maturation antigen (BCMA) chimeric antigen receptor (CAR) T cells — 0.3x10^6- 15.0x10^6 CAR+ T cells per kg of recipient bodyweight one time dose on day 0

SUMMARY:
Background:

- T cells are white blood cells that fight several cancers. One cancer therapy involves removing a persons' T cells, changing them in a lab, and then returning them to the person. Researchers want to see if this helps people with multiple myeloma.

Objective:

- To test the safety of giving anti-B-Cell Maturation Antigen T cells to people with multiple myeloma.

Eligibility:

- Adults ages 18-70 with multiple myeloma that has not responded to standard therapies.

Design:

* Participants may be screened with:
* Medical history
* Physical exam
* Blood and urine tests
* Heart tests
* Bone marrow sample
* Multiple scans and X-rays
* Participants will have apheresis. Blood is removed through a needle in an arm. T cells are removed. The rest of the blood is returned through a needle in the other arm.
* The cells will be changed in a laboratory.
* Participants will get 2 chemotherapy drugs over 3 days.
* Two days later, participants will check into the hospital. They will get an intravenous (IV) catheter in an arm or chest vein. They will get the T cells through the IV in 1 infusion.
* After this, participants will stay in the hospital for at least 9 days and stay nearby for 2 weeks. Then they will have blood tests and see a doctor.
* Participants will visit the clinic 1, 2, 3, 4, 6, and 12 months after the infusion, then every 6 months. A bone marrow sample will be taken at the 2-month visit.
* Participants blood will be collected for several years. Participants will have an annual physical at National Institutes of Health (NIH) for 5 years after the infusion. Then for 10 years they will answer health questionnaires.

DETAILED DESCRIPTION:
BACKGROUND:

* Multiple myeloma (MM) is a malignancy of plasma cells.
* MM is nearly always incurable.
* T cells can be genetically modified to express chimeric antigen receptors (CARs) that specifically target malignancy-associated antigens.
* Autologous T cells genetically modified to express CARs targeting the B-cell antigen cluster of differentiation 19 (CD19) have caused complete remissions in a small number of patients with leukemia or lymphoma. These results demonstrate that CAR-expressing T cells have anti-malignancy activity in humans.
* B-cell maturation antigen (BCMA) is a protein expressed by normal plasma cells and the malignant plasma cells of multiple myeloma.
* BCMA is not expressed by normal cells except for plasma cells and some mature B cells.
* We have constructed an anti-BCMA CAR that can specifically recognize BCMA-expressing target cells in vitro and eradicate BCMA-expressing tumors in mice.
* Anti-BCMA-CAR-expressing T cells have not been previously tested in humans.
* We hypothesize that anti-BCMA-CAR-expressing T cells will specifically eliminate

BCMA-expressing MM cells in patients

-Possible toxicities include cytokine-associated toxicities such as fever, hypotension, and neurological toxicities. Elimination of normal plasma cells and unknown toxicities are also possible.

OBJECTIVES:

Primary

-Determine the safety and feasibility of administering T cells expressing an anti- BCMA CAR to patients with MM.

Secondary

* Evaluate the in vivo persistence of anti-BCMA CAR T cells
* Assess for evidence of anti-myeloma activity by anti-BCMA CAR T cells

ELIGIBILITY

* Patients must have measurable MM defined as a serum M-protein greater than or equal to 0.4 g/dL or a urine M-protein greater than or equal to 200 mg/24 hours or an involved serum free light chain (FLC) level greater than or equal to 10 mg/dL (provided FLC ratio is abnormal) or a biopsy-proven plasmacytoma.
* Patients must have previously received at least 3 different treatment regimens for MM.
* Patients must have a normal creatinine and a normal cardiac ejection fraction.
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 -2 is required.
* Patients on any anticoagulant medications except aspirin are not eligible.
* No active infections are allowed.
* Absolute neutrophil count greater than or equal to 1000/ L, platelet count greater than or equal to 45,000/ L, hemoglobin greater than or equal to 8g/dL
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) less than or equal to 2.5-fold higher than the upper limit of normal
* At least 14 days must elapse between the time of any prior systemic treatment (including corticosteroids) and the required leukapheresis.
* At least 14 days must elapse between the time of any prior systemic treatment (including corticosteroids) and initiation of protocol treatment.
* Bone marrow plasma cells must be 30% or less of total bone marrow cells 30 days or less prior to the start of protocol treatment.
* The patient's MM will need to be assessed for BCMA expression by flow cytometry or immunohistochemistry performed at the National Institutes of Health (NIH). If unstained, paraffinembedded bone marrow or plasmacytoma sections are available from prior biopsies, these can be used to determine BCMA expression by immunohistochemistry; otherwise patients will need to come to the NIH for a bone marrow biopsy or other biopsy of a plasmacytoma to determine BCMA expression. The sample for BCMA expression can come from a biopsy obtained at any time before enrollment.

DESIGN:

* This is a phase I dose-escalation trial
* Patients will undergo leukapheresis
* T-cells obtained by leukapheresis will be genetically modified to express an anti- BCMA CAR
* Patients will receive a lymphocyte-depleting chemotherapy conditioning regimen with the intent of enhancing the activity of the infused anti-BCMA-CAR-expressing T cells.
* The chemotherapy conditioning regimen is cyclophosphamide 300 mg/m^2 daily for 3 days and fludarabine 30 mg/m^2 daily for 3 days. Fludarabine will be given on the same days as the cyclophosphamide.
* Two days after the chemotherapy ends, patients will receive an infusion of anti- BCMA-CAR-expressing T cells.
* The initial dose level of this dose-escalation trial will be 0.3x10^6 CAR+ T cells/kg of recipient bodyweight.
* The cell dose administered will be escalated until a maximum tolerated dose is determined for patients in which less than 50% of total bone marrow cells are plasma cells.

With Amendment C, all patients with 50% or greater bone marrow plasma cells will receive 3x10(6) anti-BCMA CAR T cells/kg.

* Following the T-cell infusion, there is a mandatory 9-day inpatient hospitalization to monitor for toxicity.
* Outpatient follow-up is planned for 2 weeks, and 1, 2, 3, 4, 6, 9, and 12 months after the CAR T-cell infusion.
* Repeat treatments are possible for patients with residual MM and no greater than grade 2 toxicity with an initial treatment.
* Re-enrollment will be allowed for a small number of subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

2.1.1.1 Multiple Myeloma criteria

* Clear B-cell maturation antigen (BCMA) expression must be detected on greater than 50% of malignant plasma cells from either bone marrow or a plasmacytoma by flow cytometry or immunohistochemistry. These assays must be performed at the National Institutes of Health. It is not required that the specimen used for BCMA determination comes from a sample that was obtained after the patient's most recent treatment. BCMA expression will need to be documented on the majority of malignant plasma cells at some time after the original anti-BCMA chimeric antigen receptor (CAR) T-cell infusion in all patients undergoing a second anti-BCMA CAR T-cell infusion. If paraffin embedded unstained samples of bone marrow involved with multiple myeloma (MM) or a plasmacytoma are available, these can be shipped to the National Institutes of Health (NIH) for BCMA staining, otherwise new biopsies will need to be performed for determination of BCMA expression.
* Bone marrow plasma cells must make up 30% or less of total bone marrow cells based on a bone marrow biopsy performed within 30 days of the start of protocol treatment.
* Patients must have received at least 3 different prior treatment regimens for multiple myeloma
* Patients must have measurable MM as defined by at least one of the criteria below.

  a. One or more of these abnormalities defines measurable disease:
  * Serum M-protein greater or equal to 1 g/dl (10 g/l).
  * Urine M-protein greater or equal to 200 mg/24 h.
  * Serum free light chain (FLC) assay: involved FLC level greater or equal to10 mg/dl (100 mg/l) provided serum FLC ratio is abnormal.
  * A biopsy-proven plasmacytoma
* Patients must have multiple myeloma that meets the criteria for one of the following Disease categories: (1) progressive disease or (2) relapse from Complete Remission (CR) as described in the International Uniform Response Criteria for Multiple Myeloma and as listed below.

  1. Progressive Disease (which requires 1 or more of the following)(A):

     Increase of greater than or equal to 25% from the lowest response value (nadir) in any one or more of these parameters:
     1. Serum M-component (the absolute increase must be greater than or equal to 0.5 g/dL) (B) and/or
     2. Urine M-component and/or (the absolute increase must be greater than or equal to 200 mg/24 h)
     3. Only in patients without measurable serum and urine M-protein levels; the difference between involved and uninvolved FLC levels. The absolute increase must be > 10 mg/dL.
     4. Bone marrow plasma cell percentage; the absolute percentage must be greater than or equal to 10%
* Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas (defined as 50% or greater increase in the sum of the products of the cross-diameters of target lesions)
* Development of hypercalcemia (corrected serum calcium > 11.5 mg/dL or 2.65 mmol/L) that can be attributed solely to the plasma cell proliferative disorder

  2. Relapse from complete remission (A)
* Defined as one or more of the following; must be attributable to myeloma:

  1. Reappearance of serum or urine M-protein by immunofixation or electrophoresis
  2. Development of greater than or equal to 5% plasma cells in the bone marrow
  3. Appearance of any other sign of progression (i.e., new plasmacytoma, lytic bone lesion, or hypercalcemia)

(A)All relapse and progression categories require two consecutive assessments made at any time before classification as relapse or disease progression and/or the institution of any new therapy.

(B)For progressive disease, serum M-component increases of greater than or equal to 1 gm/dL are sufficient to define progression if starting M-component is greater than or equal to 5 g/dL.

2.1.1.2 Other inclusion criteria:

* Greater than or equal to 18 years of age and less than or equal to age 73.
* Able to understand and sign the Informed Consent Document.
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0-2
* Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for four months after receiving the preparative regimen.
* Women of child bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the preparative chemotherapy on the fetus.
* Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune -competence and thus are less responsive to the experimental treatment and more susceptible to its toxicities.)
* Seronegative for hepatitis B antigen, positive hepatitis B tests can be further evaluated by confirmatory tests, and if confirmatory tests are negative, the patient can be enrolled.
* Seronegative for hepatitis C antibody unless antigen negative. If hepatitis C antibody test is positive, then patients must be tested for the presence of antigen by Reverse transcription polymerase chain reaction (RT-PCR) and be hepatitis C virus (HCV) ribonucleic acid (RNA) negative.
* Absolute neutrophil count greater than or equal to 1000/mm^3 without the support of filgrastim or other growth factors.
* Platelet count greater than or equal to 45,000/mm^3 without transfusion support
* Hemoglobin greater than 8.0 g/dl.
* Less than 5% plasma cells in the peripheral blood leukocytes
* Serum alanine transaminase (ALT) and aspartate transaminase (AST) less or equal to 2.5 times the upper limit of the institutional normal.
* Serum creatinine less than or equal to 1.3 mg/dL.
* Total bilirubin less than or equal to 2.0 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
* At least 14 days must have elapsed since any prior systemic therapy at the time the patient starts the cyclophosphamide and fludarabine conditioning regimen, and patients toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).
* Because this protocol requires collection of autologous blood cells by leukapheresis in order to prepare anti-BCMA-CAR T cells, systemic anti-myeloma therapy including systemic corticosteroid steroid therapy of greater than 5 mg/day of prednisone or equivalent dose of another corticosteroid are not allowed within 2 weeks prior to the required leukapheresis.
* Normal cardiac ejection fraction (greater than or equal to 50% by echocardiography) and no evidence of hemodynamically significant pericardial effusion as determined by an echocardiogram within 6 weeks of the start of the treatment protocol.
* Patients should not take corticosteroids including prednisone, dexamethasone or any other corticosteroid for any purpose at doses higher than 5 mg/day of prednisone or equivalent dose of another corticosteroid 2 weeks before apheresis and within 2 weeks prior to CAR T-cell infusion, and at any time after the CAR T cell infusion.

2.1.2 EXCLUSION CRITTERIA:

* Patients on any anticoagulants except aspirin are not eligible.
* Patients that require urgent therapy due to tumor mass effects or spinal cord compression.
* Patients that have active hemolytic anemia.
* Patients with second malignancies in addition to multiple myeloma are not eligible if the second malignancy has required treatment within the past 3 years or is not in complete remission. There are two exceptions to this criterion: successfully treated non-metastatic basal cell or squamous cell skin carcinoma.
* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
* Active systemic infections (defined as infections causing fevers or requiring antimicrobial treatment), active coagulation disorders or other major uncontrolled medical illnesses of the cardiovascular, respiratory, endocrine, renal, gastrointestinal, genitourinary or immune system, history of myocardial infarction, active cardiac arrhythmias, active obstructive or restrictive pulmonary disease.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Systemic corticosteroid steroid therapy of greater than 5 mg/day of prednisone or equivalent dose of another corticosteroid are not allowed within 2 weeks prior to either the required leukapheresis or the initiation of the conditioning chemotherapy regimen.
* History of severe immediate hypersensitivity reaction to any of the agents used in this study.
* History of allogeneic stem cell transplantation
* Patients with central nervous system (CNS) metastases or symptomatic CNS involvement (including cranial neuropathies or mass lesions and spinal cord compression).
* Patients with active autoimmune skin diseases such as psoriasis or other active autoimmune diseases such as rheumatoid arthritis.

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08-12 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James N Kochenderfer, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kochenderfer JN, Rosenberg SA. Treating B-cell cancer with T cells expressing anti-CD19 chimeric antigen receptors. Nat Rev Clin Oncol. 2013 May;10(5):267-76. doi: 10.1038/nrclinonc.2013.46. Epub 2013 Apr 2. PMID 23546520
- [Background] Carpenter RO, Evbuomwan MO, Pittaluga S, Rose JJ, Raffeld M, Yang S, Gress RE, Hakim FT, Kochenderfer JN. B-cell maturation antigen is a promising target for adoptive T-cell therapy of multiple myeloma. Clin Cancer Res. 2013 Apr 15;19(8):2048-60. doi: 10.1158/1078-0432.CCR-12-2422. Epub 2013 Jan 23. PMID 23344265
- [Background] Kochenderfer JN, Dudley ME, Feldman SA, Wilson WH, Spaner DE, Maric I, Stetler-Stevenson M, Phan GQ, Hughes MS, Sherry RM, Yang JC, Kammula US, Devillier L, Carpenter R, Nathan DA, Morgan RA, Laurencot C, Rosenberg SA. B-cell depletion and remissions of malignancy along with cytokine-associated toxicity in a clinical trial of anti-CD19 chimeric-antigen-receptor-transduced T cells. Blood. 2012 Mar 22;119(12):2709-20. doi: 10.1182/blood-2011-10-384388. Epub 2011 Dec 8. PMID 22160384
- [Derived] Brudno JN, Maric I, Hartman SD, Rose JJ, Wang M, Lam N, Stetler-Stevenson M, Salem D, Yuan C, Pavletic S, Kanakry JA, Ali SA, Mikkilineni L, Feldman SA, Stroncek DF, Hansen BG, Lawrence J, Patel R, Hakim F, Gress RE, Kochenderfer JN. T Cells Genetically Modified to Express an Anti-B-Cell Maturation Antigen Chimeric Antigen Receptor Cause Remissions of Poor-Prognosis Relapsed Multiple Myeloma. J Clin Oncol. 2018 Aug 1;36(22):2267-2280. doi: 10.1200/JCO.2018.77.8084. Epub 2018 May 29. PMID 29812997
- [Derived] Ali SA, Shi V, Maric I, Wang M, Stroncek DF, Rose JJ, Brudno JN, Stetler-Stevenson M, Feldman SA, Hansen BG, Fellowes VS, Hakim FT, Gress RE, Kochenderfer JN. T cells expressing an anti-B-cell maturation antigen chimeric antigen receptor cause remissions of multiple myeloma. Blood. 2016 Sep 29;128(13):1688-700. doi: 10.1182/blood-2016-04-711903. Epub 2016 Jul 13. PMID 27412889
- [Derived] Tai YT, Anderson KC. Targeting B-cell maturation antigen in multiple myeloma. Immunotherapy. 2015;7(11):1187-99. doi: 10.2217/imt.15.77. Epub 2015 Sep 15. PMID 26370838
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0168.html

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.3 x 10^6 CAR-BCMA T-cells Infused; 1 x 10^6 CAR-BCMA T-cells Infused; 3 x 10^6 CAR-BCMA T-cells Infused; 9 x 10^6 CAR-BCMA T-cells Infused: Dose Escalation with 5 dose levels based on the patients actual bodyweight
  Cyclophosphamide: 300 mg/m^2 intravenous (IV) over 30 minutes on days -5, -4, and -3
  Fludarabine: 30 mg/m^2 intravenous (IV) over 30 minutes immediately following the cyclophosphamide on day -5, -4, and -3
  Anti-B-cell maturation antigen (BCMA) chimeric antigen receptor (CAR) T cells: 0.3x10^6- 15.0x10^6 CAR+ T cells per kg of recipient bodyweight one time dose on day 0
Period: Overall Study
Arm/Group | 0.3 x 10^6 CAR-BCMA T-cells Infused | 1 x 10^6 CAR-BCMA T-cells Infused | 3 x 10^6 CAR-BCMA T-cells Infused | 9 x 10^6 CAR-BCMA T-cells Infused
Started | 3 | 3 | 5 | 19
Completed | 3 | 3 | 4 | 16
Not Completed | 0 | 0 | 1 | 3
Not completed — Patient became ineligible for treatment | 0 | 0 | 0 | 3
Not completed — Patient did not get CAR T-Cells | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.3 x 10^6 CAR-BCMA T-cells Infused | 1 x 10^6 CAR-BCMA T-cells Infused | 3 x 10^6 CAR-BCMA T-cells Infused | 9 x 10^6 CAR-BCMA T-cells Infused | Total
Number analyzed (Participants) | 3 | 3 | 5 | 19 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 5 | 17 | 28
  >=65 years | 0 | 0 | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.93 (4.87) | 54.0 (.71) | 55.76 (5.65) | 54.13 (6.86) | 56.49 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4 | 7 | 15
  Male | 0 | 2 | 1 | 12 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 4 | 4
  Not Hispanic or Latino | 3 | 3 | 5 | 14 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 2 | 5
  White | 2 | 3 | 3 | 15 | 23
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 5 | 19 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: Dose limiting toxicities are defined as follows: Grade 3 toxicities possibly or probably related to either the anti-BCMA CAR T cells or the fludarabine and cyclophosphamide chemotherapy and lasting more than 7 days. Grade 4 toxicities possibly or probably related to the study interventions.
Time Frame: After the start of treatment and up to 60 days
Population: One participant in Group 9x10(6) did not get CAR T-cells and was deemed ineligible, and 3 participants in Group 9x10(6) were found to be ineligible for treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.3 x 10^6 CAR-BCMA T-cells Infused | 1 x 10^6 CAR-BCMA T-cells Infused | 3 x 10^6 CAR-BCMA T-cells Infused | 9 x 10^6 CAR-BCMA T-cells Infused
Number analyzed (Participants) | 3 | 3 | 4 | 16
Participants
  Hypophosphatemia | 0 | 0 | 0 | 4
  Confusion | 0 | 0 | 0 | 3
  Dyspnea (intubated) | 0 | 0 | 0 | 4
  Ejection fraction decreased | 0 | 0 | 0 | 4
  Encephalopathy | 0 | 0 | 0 | 3
  Hypoxia | 0 | 0 | 0 | 3
  Acute kidney injury (CVVH) | 0 | 0 | 0 | 4
  Sepsis (Staph Aureus) | 0 | 0 | 0 | 4
  Muscle weakness lower limbs | 0 | 0 | 0 | 3
  Muscle weakness upper limbs | 0 | 0 | 0 | 3
  Platelet count decreased | 0 | 0 | 0 | 3
  Neutrophil count decreased | 0 | 0 | 0 | 4
  Acute kidney injury | 0 | 0 | 0 | 3
  Hypotension | 0 | 0 | 0 | 4
  CPK increased | 0 | 0 | 0 | 4
  Musculoskeletal/connective tissue disorders-Rhabd. | 0 | 0 | 0 | 3

2. Primary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approx. 3 mos and 7 days for DL 0.3 x 10^6 CAR + T cells, 4 mos and 4 days for 1.0 x 10^6 CAR + T cells, 9 mos and 13 days for 3.0 x 10^6 CAR + T cells, and 48 mos and 12 days for 9.0 x 10^6 CAR + T cells.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 0.3 x 10^6 CAR-BCMA T-cells Infused | 1 x 10^6 CAR-BCMA T-cells Infused | 3 x 10^6 CAR-BCMA T-cells Infused | 9 x 10^6 CAR-BCMA T-cells Infused
Number analyzed (Participants) | 3 | 3 | 4 | 16
Participants | 3 | 3 | 4 | 16

3. Secondary Outcome: Number of Participants With Best Response
Description: Best response was assessed by the International Myeloma Working Group response criteria. Partial Remission (PR) is 50% or greater reduction of serum M-protein and 90% or greater reduction in 24-h urinary M-protein. Progressive Disease (PD) is increases of greater or equal to 25% from the lowest post-treatment (nadir) value in serum M-component or urine component or percentage of bone marrow plasma cells. Definite development of new bone lesions or new plasmacytoma. Very Good Partial Remission (VGPR) is serum and urine M-protein detectable by immunofixation but not on electrophoresis. Stringent Complete Remission (sCR) is normal free light chain ratio and absence of clonal cells in bone marrow by immunohistochemistry. Complete Remission is negative immunofixation on the serum and urine. Stable Disease (SD) is not meeting criteria for CR, VGPR, PR or PD.
Time Frame: From start of treatment up to 84 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 0.3 x 10^6 CAR-BCMA T-cells Infused | 1 x 10^6 CAR-BCMA T-cells Infused | 3 x 10^6 CAR-BCMA T-cells Infused | 9 x 10^6 CAR-BCMA T-cells Infused
Number analyzed (Participants) | 3 | 3 | 4 | 16
Participants
  Partial Remission | 1 | 0 | 0 | 4
  Stable Disease | 2 | 3 | 3 | 2
  Very Good Partial Remission | 0 | 0 | 1 | 6
  Complete Remission | 0 | 0 | 0 | 1
  Stringent Complete Remission | 0 | 0 | 0 | 2
  Progressive Disease | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 3 months and 7 days for dose level 0.3 x 10^6 CAR + T cells, 4 months and 4 days for 1.0 x 10^6 CAR + T cells, 9 months and 13 days for 3.0 x 10^6 CAR + T cells, and 48 months and 12 days for 9.0 x 10^6 CAR + T cells.
Description: One participant in Group 9x10(6) did not get CAR T-cells and was deemed ineligible, and 3 participants in Group 9x10(6) were found to be ineligible for treatment.
Arm/Group | 0.3 x 10^6 CAR-BCMA T-cells Infused | 1 x 10^6 CAR-BCMA T-cells Infused | 3 x 10^6 CAR-BCMA T-cells Infused | 9 x 10^6 CAR-BCMA T-cells Infused
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/4 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 1/4 | 11/16
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.3 x 10^6 CAR-BCMA T-cells Infused (N=3) | 1 x 10^6 CAR-BCMA T-cells Infused (N=3) | 3 x 10^6 CAR-BCMA T-cells Infused (N=4) | 9 x 10^6 CAR-BCMA T-cells Infused (N=16)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
White blood cell decreased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (7)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Cardiac troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Infections and infestations - Other, CMV viremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, Salmonella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Rhabdomyalysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.3 x 10^6 CAR-BCMA T-cells Infused (N=3) | 1 x 10^6 CAR-BCMA T-cells Infused (N=3) | 3 x 10^6 CAR-BCMA T-cells Infused (N=4) | 9 x 10^6 CAR-BCMA T-cells Infused (N=16)
Anemia (Blood and lymphatic system disorders) | 3 (4) | 2 (2) | 4 (7) | 13 (42)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 7 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 2 (5) | 14 (59)
Lymphocyte count decreased (Investigations) | 3 (9) | 3 (7) | 4 (10) | 14 (49)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 12 (15)
Neutrophil count decreased (Investigations) | 3 (13) | 3 (12) | 4 (14) | 16 (68)
Platelet count decreased (Investigations) | 2 (5) | 1 (1) | 2 (5) | 11 (58)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 8 (11)
White blood cell decreased (Investigations) | 3 (14) | 3 (14) | 4 (18) | 16 (69)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 7 (9)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Fever (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 15 (36)
Hyponatremia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CPK increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (11)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 15 (31)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acidosis (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alkalosis (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (6)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 6 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (18)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (9)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, Clostridium difficile stool (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 11 (14)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Basal cell carcinoma removal (face and upper back)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Basal cell carcinoma (L base of neck)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Basal cell carcinoma (L cheek)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Basal cell carcinoma (upper back)
Infections and infestations - Other, Clostridium difficile (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/67/NCT02215967/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT02215967/ICF_001.pdf